CLINICAL TRIAL: NCT02998554
Title: A Phase 3, Multi-center, Randomized, Double-Masked Study to Evaluate the Clinical Efficacy and Safety of SHP640 (PVP-Iodine 0.6% and Dexamethasone 0.1%) Ophthalmic Suspension Compared to Placebo in the Treatment of Adenoviral Conjunctivitis
Brief Title: Treatment of Adenoviral Conjunctivitis With SHP640 Compared to Placebo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision, unrelated to safety
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP640-302; 2016-002440-16 (EudraCT Number)
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Results first posted 2020-05-29 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Adenoviral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHP640 (Experimental): Participants instructed to instill 1 drop of SHP640 (Povidone-iodine [PVP-I] 0.6 percent [%] and Dexamethasone 0.1%) ophthalmic suspension in each eye 4 times daily (QID) (with a minimum of 2 hours between doses) for 7 days.
  Interventions: Drug: SHP640
- Placebo (Placebo Comparator): Participants instructed to instill 1 drop of placebo ophthalmic solution in each eye QID for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHP640 — Instill 1 drop of SHP640 (PVP-I 0.6% and Dexamethasone 0.1%) ophthalmic suspension in each eye 4 times daily (QID) (with a minimum of 2 hours between doses) for 7 days.
  Arms: SHP640
Drug: Placebo — Instill 1 drop of placebo ophthalmic solution in each eye QID for 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if an investigational treatment is effective compared with placebo in the treatment of adults and children with adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria

1. An understanding, ability, and willingness to fully comply with study procedures and restrictions (by the parent(s), guardian, or legally authorized representative, if applicable).
2. Ability to voluntarily provide written, signed, and dated (personally or via a parent(s), guardian, or legally-authorized representative(s) informed consent (and assent, if applicable) to participate in the study.
3. Participants of any age at Visit 1 (Note: Participants less than (<) 3 months of age at Visit 1 must have been full-term, that is greater than or equal to (>=) 37 weeks gestational age at birth).
4. Meet at least 1 of the 2 criteria below: a. Have a positive AdenoPlus® test at Visit 1 in at least 1 eye; b. Have at least 2 of the following 5 criteria, based upon medical history and examination: i. Symptoms within the past 7 days consistent with acute upper respiratory tract infection (example: sore throat, cough, rhinorrhea, etc); ii. Contact within the past 7 days with family members or other individuals with recent onset of symptoms consistent with conjunctivitis; iii. Acute onset within the past 4 days of 1 or more of the following ocular symptoms: burning/irritation, foreign body sensation, light sensitivity; iv. Enlarged periauricular lymph node(s); v. Presence of follicles on tarsal conjunctiva.

   Note: If the participant only meets Inclusion Criterion 4a (a positive AdenoPlus test in at least 1 eye), then the same eye must meet Inclusion Criterion 5.
5. Have a clinical diagnosis of suspected adenoviral conjunctivitis in at least 1 eye confirmed by the presence of the following minimal clinical signs and symptoms in that same eye: Report presence of signs and/or symptoms of adenoviral conjunctivitis for less than or equal to (<=) 4 days prior to Visit 1; Bulbar conjunctival injection: a grade of >=1 on 0-4 scale of Bulbar Conjunctival Injection Scale; Watery conjunctival discharge: a grade of >=1 (mild) on a 0-3 Watery Conjunctival Discharge Scale.
6. Be willing to discontinue contact lens wear for the duration of the study.
7. Have a Best Corrected Visual Acuity (BCVA) of 0.60 logMAR or better in each eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. BCVA will be assessed by an age appropriate method in accordance with the American Academy of Pediatrics (AAP) Policy Statement for Visual System Assessment in Infants, Children, and Young Adults by Pediatricians. The policy statement recommends formal vision screening can begin at 3 years of age. VA measurements for children under the age of 3 will be done at the discretion of the investigator. If not done, child should be able to fixate on and follow a moving object, except participants < 2 months of age who have not yet developed this ability. Participants < 2 months will be enrolled at the discretion of the investigator.
8. Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Exclusion Criteria

1. Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments, per investigator's discretion.
2. Current or relevant history of physical or psychiatric illness, any medical disorder that may make the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
3. Have known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.
4. Prior enrollment in a FST-100 or SHP640 clinical study.
5. Participants who are employees, or immediate family members of employees (who are directly related to study conduct), at the investigational site.
6. Have a history of ocular surgical intervention within <= 6 months prior to Visit 1 or planned for the period of the study.
7. Have a preplanned overnight hospitalization during the period of the study.
8. Have presence of any intraocular, corneal, or conjunctival ocular inflammation (example: uveitis, iritis, ulcerative keratitis, chronic blepharoconjunctivitis), other than adenoviral conjunctivitis.
9. Have presence of corneal subepithelial infiltrates at Visit 1.
10. Have active or history of ocular herpes.
11. Have at enrollment or within <= 30 days of Visit 1, a clinical presentation more consistent with the diagnosis of non-infectious conjunctivitis (except presumed seasonal/perennial allergic conjunctivitis) or non-adenoviral ocular infection (example: bacterial, fungal, acanthamoebal, or other parasitic).

    Note: History or concomitant presence of presumed seasonal or perennial allergic conjunctivitis signs/symptoms is not exclusionary.
12. Neonates or infants (that is (ie,) participants < 12 months of age) who have suspected or confirmed (based on the result of any test conducted prior to screening) conjunctivitis of gonococcal, chlamydial, herpetic or chemical origin.
13. Neonates or infants (ie, participants < 12 months of age) whose birth mothers had any sexually transmitted disease within 1 month of delivery or any history of genital herpes.
14. Presence of nasolacrimal duct obstruction at Visit 1 (Day 1).
15. Presence of any significant ophthalmic condition (example: retinopathy of prematurity, congenital cataract, congenital glaucoma) or other congenital disorder with ophthalmic involvement that could affect study variables.
16. Be a known intraocular pressure (IOP) steroid responder, have a known history or current diagnosis of glaucoma, or be a glaucoma suspect.
17. Have any known clinically significant optic nerve defects.
18. Have a history of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome; presence of corneal epithelial defect or any significant corneal opacity at Visit 1.
19. Presence of significant, active condition in the posterior segment which requires invasive treatment (example: intravitreal treatment with VEGF inhibitors or corticosteroids) and may progress during the study participation period.
20. Have used any topical ocular or systemic anti-virals or antibiotics within <= 7 days of enrollment.
21. Have used any topical ocular NSAIDs within <= 1 day of enrollment.
22. Have used any topical ophthalmic steroids in the last <= 14 days.
23. Have used any systemic corticosteroid agents within <= 14 days of Day 1. Stable (initiated >= 30 days prior to enrollment) use of inhaled and nasal corticosteroids is allowed, given no anticipated change in dose for the duration of the study. Topical dermal steroids are allowed except in the peri-ocular area.
24. Have used non-corticosteroid immunosuppressive agents within <= 14 days of Day 1.
25. Have used any topical ophthalmic products, including tear substitutes, and over-the-counter preparations such as lid scrubs, within 2 hours of Visit 1 and be unable to discontinue all topical ophthalmic products for the duration of the study. Use of hot or cold compresses is also not permitted during the study.
26. Have any significant ocular disease (example: Sjogren's syndrome) or any uncontrolled systemic disease or debilitating disease (example: cardiovascular disease, hypertension, sexually transmitted diseases/infections, diabetes or cystic fibrosis), that may affect the study parameters, per investigator's discretion.
27. Any known history of immunodeficiency disorder or known active conditions predisposing to immunodeficiency, such as human immunodeficiency virus, hepatitis B or C, evidence of active hepatitis A (antihepatitis A virus immunoglobulin M), or organ or bone marrow transplantation.
28. Within 30 days prior to the first dose of investigational product: Have used an investigational product or device, or Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- United States (29):
  - Lugene Eye Institute Inc, Glendale, California
  - University of Southern California, Los Angeles, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Danbury Eye Physicians and Surgeons, Danbury, Connecticut
  - Bruce A. Segal, MD, PA, Delray Beach, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Inc., Largo, Florida
  - South Florida Research Center Inc., Miami, Florida
  - International Research Center, Tampa, Florida
  - Saltzer Medical Group, Nampa, Idaho
  - Sabates Eye Centers, Leawood, Kansas
  - Physicians to Children & Adolescents, Bardstown, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Shire Call Center, Lexington, Massachusetts
  - Silverstein Eye Centers, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Wellish Vision Institute, Las Vegas, Nevada
  - Fichte, Endl and Elmer Eyecare, Niagara Falls, New York
  - Apex Eye Kenwood, Cincinnati, Ohio
  - Cleveland Eye Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Eyeland Vision, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Sun Research Institute, LLC, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Piedmont Eye Center, Inc., Lynchburg, Virginia
- Puerto Rico (2):
  - Emanuelli Research & Development Center, LLC, Arecibo
  - University Of Puerto Rico, School of Medicine, Carolina

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 30 centers in the United States and Puerto Rico between 28 March 2017 (first participant first visit) and 16 May 2019 (last participant last visit).
Pre-assignment Details: A total of 156 participants were randomized and received the treatment. Out of them, 134 participants completed the study.
Groups:
- SHP640: Participants administered one drop of SHP640 (Povidone-iodine [PVP-I] 0.6 percent [%] and Dexamethasone 0.1%) ophthalmic suspension in each eye 4 times daily (QID) for 7 days.
- Placebo: Participants administered one drop of placebo ophthalmic solution in each eye QID for 7 days.
Period: Overall Study
Arm/Group | SHP640 | Placebo
Started | 79 | 77
Completed | 68 | 66
Not Completed | 11 | 11
Not completed — Adverse Event | 8 | 3
Not completed — Protocol deviation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all screened participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | SHP640 | Placebo | Total
Number analyzed (Participants) | 79 | 77 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (21.57) | 41.3 (21.21) | 41.9 (21.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 100
  Male | 32 | 24 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 19 | 29
  Not Hispanic or Latino | 68 | 58 | 126
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 64 | 68 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Resolution on Day 6
Description: Clinical resolution of adenoviral conjunctivitis was defined as the absence (score = 0) of bulbar conjunctival injection and watery conjunctival discharge in the study eye. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her cell culture-immunofluorescence assay (CC-IFA) results at baseline. Higher scores represented worse symptoms for both scales. Percentage of participants with clinical resolution on Day 6 was reported.
Time Frame: Day 6
Population: Modified Intent to Treat (mITT) population consisted of a subset of the ITT Population who received at least one dose of investigational product and has a positive CC-IFA adenovirus test at baseline in the study eye. Here, the number of participants analyzed refer to the participants evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 9 | 10
Percentage of participants | 11.1 | 20.0

2. Secondary Outcome: Percentage of Participants With Adenoviral Eradication on Day 6
Description: Adenoviral eradication for the study eye was defined as negative CC-IFA in that eye. The CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline. Percentage of participants with adenoviral eradication on Day 6 was reported.
Time Frame: Day 6
Population: mITT population consisted of a subset of the ITT Population who received at least one dose of investigational product and has a positive CC-IFA adenovirus test at baseline in the study eye. Here, the number of participants analyzed refer to the participants evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 9 | 10
Percentage of participants | 33.3 | 70.0

3. Secondary Outcome: Absolute Change and Change From Baseline in Adenovirus Viral Titer on Day 6 and 8
Description: Adenovirus viral titer was assessed by quantitative polymerase chain reaction (qPCR) in the study eye. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline.
Time Frame: Day 6 and 8
Population: The study was terminated as the sponsor discontinued the SHP640 clinical development with reason unrelated to safety. Hence, for this outcome measure, the planned data collection and analysis was not performed.
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Adenoviral Eradication on Day 3, 8 and 12/Early Termination (ET)
Description: Adenoviral eradication for the study eye was defined as negative CC-IFA in that eye. CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline. Percentage of participants with adenoviral eradication on Day 3, 8 and 12/ET was reported.
Time Frame: Day 3, 8 and 12/ET
Population: mITT population consisted of a subset of the ITT Population who received at least one dose of investigational product and has a positive CC-IFA adenovirus test at baseline in the study eye. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specific time point.
Measure: Number; unit: Percentage of participants
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 9 | 12
Percentage of participants
  Day 3 | 11.1 | 16.7
  Day 8: number analyzed (Participants) | 7 | 9
  Day 8 | 71.4 | 66.7
  Day 12/ET: number analyzed (Participants) | 9 | 11
  Day 12/ET | 77.8 | 100

5. Secondary Outcome: Percentage of Participants With Clinical Resolution on Day 3, 8 and 12/Early Termination (ET)
Description: Clinical resolution of adenoviral conjunctivitis was defined as the absence (score = 0) of bulbar conjunctival injection and watery conjunctival discharge in the study eye. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her cell culture-immunofluorescence assay (CC-IFA) results at baseline. Higher scores represented worse symptoms for both scales. Percentage of participants with clinical resolution on Day 3, 8 and 12/ET was reported.
Time Frame: Day 3, 8 and 12/ET
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 9 | 12
Percentage of participants
  Day 3 | 11.1 | 0
  Day 8: number analyzed (Participants) | 7 | 9
  Day 8 | 14.3 | 44.4
  Day 12/ET | 33.3 | 50.0

6. Secondary Outcome: Number of Participants With Individual Clinical Signs Score at Day 3, 6, 8 and 12/Early Termination (ET)
Description: Individual clinical signs scores for bulbar conjunctival injection and watery conjunctival discharge in the study eye were reported. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). Higher score represented worse symptoms for both scores. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 3
Groups:
- SHP640: Participants received 1 drop of SHP640 (Povidone-iodine [PVP-I] 0.6 percent [%] and Dexamethasone 0.1%) ophthalmic suspension in each eye 4 times daily (QID) (with a minimum of 2 hours between doses) for 7 days.
- Placebo: Participants received 1 drop of placebo matched to SHP640 ophthalmic solution in each eye QID for 7 days.
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Global Clinical Score at Day 3, 6, 8 and 12/Early Termination (ET)
Description: Global clinical score was the sum of bulbar conjunctival injection and watery conjunctival discharge in the study eye. Score range from 0 to 7 and higher scores represented worse symptoms. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 3
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With Modified Clinical Resolution at Day 3, 6, 8 and 12/Early Termination (ET)
Description: Modified clinical resolution was defined as a global clinical score of 0 or 1 in the study eye. Global clinical score was the sum of bulbar conjunctival injection and watery conjunctival discharge. Score range from 0 to 7 and higher scores represent worse symptoms.The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 3
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Expanded Clinical Resolution at Day 3, 6, 8 and 12/Early Termination (ET)
Description: Expanded clinical resolution was defined as a global clinical score of 0, 1, or 2 with neither injection nor discharge having a score of 2 in the study eye. Global clinical score was the sum of bulbar conjunctival injection and watery conjunctival discharge. Score range from 0 to 7 and higher scores represent worse symptoms. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 3
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants With Cross-Over Infection at Day 3, 6, 8 and 12/Early Termination (ET)
Description: Cross-over infection to a participant's fellow eye for participants with only 1 infected eye at baseline was reported. The CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 3
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Clinical Resolution on Day 3, 6, 8 and 12/Early Termination (ET)
Description: Time to clinical resolution was reported based on the assessments in the study eye.The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores, as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 3
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any unfavorable and unintended sign, symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. Treatment-Emergent Adverse Events (TEAEs) were defined as those adverse events that occurred after the first dose of investigational product.
Time Frame: From start of study drug administration up to Day 13
Population: Safety Population consisted of all screened participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | Placebo
Number analyzed (Participants) | 79 | 77
Participants | 28 | 17

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 13
Arm/Group | SHP640 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/77
Other Adverse Events (participants affected / at risk) | 20/79 | 8/77
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP640 (N=79) | Placebo (N=77)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0)
Corneal infiltrates (Eye disorders) | 2 (2) | 2 (2)
Dry eye (Eye disorders) | 6 (6) | 2 (2)
Erythema of eyelid (Eye disorders) | 0 (0) | 2 (2)
Instillation site pain (General disorders) | 6 (6) | 3 (3)
Conjunctivitis (Infections and infestations) | 5 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated as the sponsor discontinued the SHP640 clinical development with reason unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT02998554/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT02998554/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT02998554/Prot_002.pdf
  • Study Protocol: Amendment 3 (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02998554/Prot_003.pdf
  • Study Protocol: Amendment 4 (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT02998554/Prot_004.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT02998554/SAP_005.pdf